CLINICAL TRIAL: NCT03884829
Title: A Phase I Pharmacologic Study of CYC140, a Polo-like Kinase 1 Inhibitor, in Patients with Advanced Leukemias or Myelodysplastic Syndromes
Brief Title: A Phase I Study of CYC140, a PLK-1 Inhibitor, in Advanced Leukemias or MDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Switch to oral formulation of CYC140 (plogosertib)
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC140-01
Record Dates: First submitted 2018-10-28; First posted 2019-03-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AML, Adult; Myelodysplastic Syndromes; ALL, Adult; CML, Refractory; CLL, Refractory
Keywords: AML, ALL, CLL, CML, MDS, advanced leukemias, leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Intervention Model Description: One to three patients will be entered at a given dose level of CYC140. During the first cycle, all patients will be evaluated for DLTs. If DLT occurs, additional patients (up to 3) will be dosed at that dose. If no additional DLTs observed, dose escalation will continue per protocol. If a DLT does occur, dose escalation will be stopped. At least 6 patients will be treated at the RD to confirm its tolerability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CYC140 single agent (Experimental): CYC140 will be administered as a single agent on Day 1 and Day 8 of each 3 week cycle
  Interventions: Drug: CYC140

INTERVENTIONS:
Drug: CYC140 — CYC140 single agent

SUMMARY:
A Phase I Pharmacologic Study of CYC140, a polo-like kinase 1 inhibitor, in Patients with Advanced Leukemias or Myelodysplastic Syndromes

DETAILED DESCRIPTION:
This is a First in Human, open-label, single arm, dose escalation study in patients with advanced leukemias or myelodysplastic syndromes. Patients will receive CYC140 as a 1 hr infusion once a week for 2 weeks followed by 1 week of rest on an outpatient basis. One treatment cycle is 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory advanced leukemias or MDS
* ECOG 0-2
* Adequate renal function
* Adequate liver function
* ≥ 2 weeks from prior chemotherapy, radiation therapy or major surgery
* ≥ 4 weeks from other investigational anticancer therapy
* Agree to practice effective contraception

Exclusion Criteria:

* Known CNS involvement by leukemia
* Currently receiving radiotherapy, biological therapy, or any other investigational agents
* Uncontrolled intercurrent illness
* Pregnant or lactating
* Known to be HIV-positive
* Known active hepatitis B and/ or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Number of Patients who experience dose -limiting toxicity (DLT) | At end of cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Pharmacokinetic measurement - area under the curve (AUC) | At the end of cycle 1 (each cycle is 21 days)
  plasma drug exposure area under the curve (AUC)

OTHER OUTCOMES:
Anti-tumor activity | First dose of CYC140 to 4 weeks after the last dose of CYC140
  complete remission, partial remission

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No